CLINICAL TRIAL: NCT07347834
Title: TRIOCOL - The Study of Continued Advanced Medical Therapy or Colectomy in Patients With Ulcerative Colitis
Acronym: TRIOCOL
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other); University Hospital, Linkoeping (Other); Linkoeping University (Other Government)
Responsible Party: Sponsor
Other Study IDs: KI 4-3290/2024
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative colitis; Advanced medical therapy; Colectomy; Health related quality of life; Shared decision-making
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Contunued advanced medical therapy: If the patient chooses continued medical therapy, the gastroenterologist evaluates the patient for a new line of AMT in accordance with clinical practice. The study period starts on the date of initiation of the new drug.
- Colectomy: If the patient chooses colectomy the surgeon will inform the patient further, schedule the surgery, and if needed commence with preoperative optimization in accordance with standard clinical practice. The study period starts at the date of surgery.

SUMMARY:
Ulcerative colitis is an inflammatory disease affecting the rectum and colon, most commonly presenting in late adolescence or early adulthood. The primary treatment approach is pharmacological. Over the past two decades, there has been significant progress in the development of so-called advanced medical therapies, and new drugs in this category continue to emerge. These medications are highly effective for many patients, but not for all. If the first advanced therapy fails or is not tolerated, patients may switch to a second, third, or subsequent drugs. Unfortunately, the likelihood of success decreases with each additional line of therapy.

An alternative is surgery, specifically colectomy, which is a potentially curative treatment but may have a major impact on the individual. The overall objective of the study is to evaluate quality of life, functional outcomes, and patient satisfaction among those who choose continued medical therapy, compared to those who undergo colectomy, after at least two failed advanced medical therapies. Before making their treatment decision and enrolling in the study, patients will receive standardized information about all treatment options from a gastroenterologist and a colorectal surgeon. The aim is that the results of this study will provide valuable insights to better guide future patients with ulcerative colitis in choosing between continued advanced medical therapy and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with UC with active disease
* failed at least two lines of advanced medical therapies
* are eligible for both continued AMT and colectomy

Exclusion Criteria:

* diagnostic uncertainty
* diagnosis of impaired cognitive function
* non-domestic and non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all adult patients (≥18 years) with UC with active disease, at any of the participating centres, who have failed at least two lines of AMTs, and are eligible for both continued AMT and colectomy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
HRQoL at six months | Primary endpoint evaluated six months after enrollement.
  The patients will be evaluated with electronically distributed questionnaires at six months. The primary endpoint, health related quality of life (HRQOL), will be evaluated with 36-Item Short Form Survey (SF-36). Range 0-100. Higher number indicated better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nordenvall, Ass. professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Legal agreements will be set up between all sites that will contribute data to the study.
Supporting Information: Study Protocol, SAP